CLINICAL TRIAL: NCT04173754
Title: Observational Study on Effectiveness of MSAT(Motion Style Acupuncture Treatment) for Patients With ROM(Range of Motion) Limitation of the Shoulders Due to the Shoulder Diseases
Brief Title: The Effectiveness of MSAT for Patients With ROM Limitation of the Shoulders
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2019-10
Record Dates: First submitted 2019-11-14; First posted 2019-11-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Shoulder Joint Disorder
Keywords: Shoulder joints; ROM; Shoulder disorder; MSAT; Motion Style Acupuncture Treatment; Shoulder pains
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MSAT Group: The MSAT group who are treated with korean medical treatment including MSAT will be evaluated on first, second, third visit and 2weeks after baseline. And the patients will receive telephone inquires after 3months from the baseline.
  The Korean medical treatment includes acupuncture, chuna, pharmaco-acupuncture and Korean herbal medicine.
  Interventions: Procedure: Motion Style Acupuncture Treatment(MSAT)
- Control Group: The control group who are treated with Korean medical treatment not including MSAT will be evaluated on first, second, third visit and 2weeks after baseline. And the patients will receive telephone inquires after 3months from the baseline.
  The Korean medical treatment includes acupuncture, chuna, pharmaco-acupuncture and Korean herbal medicine.

INTERVENTIONS:
Procedure: Motion Style Acupuncture Treatment(MSAT) — Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation
  Groups: MSAT Group

SUMMARY:
This study is a prospective, case-control observational trial. The investigators will compare the MSAT group to the control group to analyze the effectiveness of shoulder MSAT.

DETAILED DESCRIPTION:
Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation. This treatment is known to relieve the pain and increase the range of motion(ROM). However, there has been no specific value for the effect of this treatment.

Therefore, The investigators conducted observational trial to analyze the effectiveness of shoulder MSAT. From July 2019, The investigators will collect 80 patients with ROM limitation on both or each shoulder and who are suffering from shoulder pain with the numeric rating scale(NRS) over 4.

The investigators will compare pain, dysfunction, quality of life and satisfaction of patients who are treated with Korean medical treatment including MSAT and patients who are treated with Korean medical treatment not including MSAT.

For these two groups, The investigators will compare Range Of Motion(ROM), NRS(Numeric Rating Scale), Visual Analogue Scale(VAS), Shoulder Pain and Disability Index(SPADI), Patient Global Impression of Change (PGIC) and EuroQol 5-Dimension (EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than one ROM limitation(Abduction 180˚, Adduction 45˚, Flexion 180˚, Extension 45˚, Int. rot 80˚, Ext. rot 80˚) on both or each shoulder.
* Patients with NRS ≥ 4 for shoulder pain
* Patients aged 19-70 years on the date they sign the consent form.
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients who have been diagnosed with a severe disease that may cause ROM limitation of shoulder or shoulder pain,
* Patients with progressive neurological deficit or with serious neurological symptoms caused by spinal cord compression.
* Patients who visited a hospital in pain caused by a traffic accident.
* Patients with a severe mental illness.
* Patients who are difficult to complete the research participation agreement

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated in Haeundae Jaseng Korean Medicine Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Shoulder mobility on the Shoulder ROM | At within 2 weeks
  Shoulder ROM was measured in six directions (Flexion, Extension, Abduction, Adduction, Right rotation, Left rotation) with goniometer.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) of shoulder pain | At screening, baseline, 2 weeks, 3 months, and through study completion, an average of 3 month
  The extent of shoulder pain and discomfort was assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their shoulder pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual Analogue Scale (VAS) of shoulder pain | At screening, baseline, 2 weeks and through study completion, an average of 3 month
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Shoulder Pain and Disability Index(SPADI) questionnaire of shoulder pain and disability | At baseline, 2 weeks, 3 months
  SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.
Patient Global Impression of Change (PGIC) | At baseline, 2 weeks, 3 months
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
EuroQol 5-Dimension (EQ-5D-5L) | At baseline, 2 weeks, 3 months
  The EQ-5D-5L is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, The investigators will use the Korean version of the EQ-5D-5L, which has been demonstrated to be valid.
Adverse events(AE) | Through study completion, an average of 3 month
  Adverse events(AE) Physicians will monitor and record any unexpected or unintended patient reaction to integrative korean medicine at each visit. Adverse events (AEs) associated with integrative korean medicine will include, but not be limited to, AEs anticipated from previous reports of korean medicine, and will stay open to all possibilities taking into consideration other potential, unknown AEs.
Shoulder mobility on the Shoulder ROM | At screening, baseline, 2 weeks, 3 months and through study completion, an average of 3 month
  Shoulder ROM was measured in six directions (Flexion, Extension, Abduction, Adduction, Right rotation, Left rotation) with goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Study Chair — Jaseng Medical Foundation
Locations (1):
- Haeundae Jaseng Hospital of Korean Medicine, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided